CLINICAL TRIAL: NCT05215691
Title: TAPA Block Versus Conventional Analgesia Methods on Cognitive Functions and Postoperative Opioid Consumption in Major Abdominal Surgery
Brief Title: Outcomes of Thoracoabdominal Nerve Block Through Perichondrial Approach* on Postoperative Cognitive Functions
Acronym: TAPA
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Guldeniz Argun, associate professor, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2021-04/1098
Record Dates: First submitted 2021-12-03; First posted 2022-01-31 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Cognition
Keywords: TAPA block, opioid consumption, cognitive functions
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I (n=45, TAPA): The patients who received TAPA block for postoperative analgesia are named as a Group I ( n=45). The TAPA block is performed at the rib margin where the 9th and 10th ribs meet. A linear transducer is placed at the costochondral angle in the sagittal plane. It is carried out by injecting 20 ml of Bupivacaine %0.200 between the upper and lower surface of the chondrium. All patients receive IV PCA with morphine 0.5 mg/ml.
  Interventions: Procedure: Group I: TAPA block
- Group II (n=45, IV opioid): The patients who did not prefer the block and preferred intravenous patient-controlled analgesia (PCA) are named as Group II (n=45). IV PCA is prepared with morphine 0.5 mg/ml.
  Interventions: Procedure: Group II: IV Morphine

INTERVENTIONS:
Procedure: Group I: TAPA block — Postoperative analgesia will be provided with peripheral nerve block (TAPA)
  Other Names: thoracoabdominal block perichondral appearance
  Groups: Group I (n=45, TAPA)
Procedure: Group II: IV Morphine — Postoperative analgesia will be provided with opioids
  Other Names: intravenous morphine group
  Groups: Group II (n=45, IV opioid)

SUMMARY:
It was planned to compare the opioid consumption and cognitive functions in the postoperative period of patients who received TAPA block for postoperative analgesia and patients who did not prefer the block and who preferred intravenous patient-controlled analgesia (PCA) with opioids. Both the surgery applied and the drugs used in anesthesia can cause changes in cognitive functions by affecting the inflammatory process. It is thought that if the patients' pain can be relieved sufficiently in the postoperative period with TAPA block, the consumption of opioids used will be less and their cognitive functions will be less affected.

DETAILED DESCRIPTION:
Postoperative pain management after major surgical operations is a very important issue. Features such as waking up without pain, early recovery from anesthesia, not suppressing respiration by the drugs used for postoperative pain treatment, not delaying recovery from anesthesia, not having unwanted side effects, and not delaying discharge from the intensive care unit are the desired features of postoperative pain management. A wide variety of drug therapy modalities are available for this purpose. However, peripheral nerve blocks are widely used to minimize undesirable effects of drug therapy. TAP block (trans abdominal plane block) has been used for this purpose since ancient times. TAPA block (thoracoabdominal block with perichondral approach) is a newly developed plane block and was developed to obtain higher level block with a single injection. In this study, we planned to compare the recovery times from anesthesia, postoperative pain scores, opioid consumption, and cognitive functions of patients who underwent TAPA block for postoperative pain treatment and patients who were not preferred to TAPA block and were planned for pain treatment with conventional methods, whether these treatments affected or not.

Neuropsychological dysfunction is a frequently encountered condition after surgery. Postoperative cognitive dysfunction can affect various cognitive functions such as attention, memory, and information processing speed. The most notable symptoms are memory deficits and decreased ability to cope with intellectual difficulties. It has been stated that postoperative cognitive dysfunction depends on advanced age, duration of anesthesia, development of complications, pre-existing cognitive disorders, and education level.

In a study, it was reported that the incidence of postoperative cognitive dysfunction in patients aged around 60 years who underwent major noncardiac surgery was 25.8% after 1 week and 9.9% after 3 months.

In the literature, it has been mentioned that inflammatory processes that occur as a result of surgical trauma and subsequent complications play a role in cognitive dysfunction. Normal cognitive functions can be maintained in low-level inflammatory processes, while very high-level proinflammatory factors can significantly affect cognitive functions.

Traditional lateral TAP block is performed on the midaxillary line between the iliac crest and subcostal. With this approach, with cadaveric dye injection, T11 was shown to be maintained and T12 was maintained 100% time, L1 93% time and T10 50% time. The lateral TAP block reached a dermatome high enough to benefit the patient after open cholecystectomy.

The TAPA block is performed at the rib margin where the 9th and 10th ribs meet. A linear transducer is placed at the costochondral angle in the sagittal plane. It is carried out by injecting 20 ml of drug between the upper and lower surface of the chondrium. The authors state that TAPA block provides analgesia to T5-T12. They hypothesize that the TAPA block numbs both the lateral cutaneous branch and the anterior region.

Although the standardized mini-mental test is not a definitive diagnostic test, it is used by clinicians as an auxiliary test to measure the degree of cognitive deterioration of patients.

We planned this study to compare the recovery times from anesthesia, postoperative pain scores, opioid consumption, and cognitive functions of patients who underwent TAPA block for postoperative pain management and patients who were not preferred TAPA block and were planned for pain treatment with conventional methods, whether these treatments were affected or not.

ELIGIBILITY:
Inclusion Criteria:

1. patients who will undergo major abdominoplasty,
2. over the age of 18,
3. under the age of 85,
4. patients who has ASA (American Society of Anesthesiologists) II and ASA III criteria

Exclusion Criteria:

1. younger than 18 years old, over 85 years old,
2. Having a history of cerebrovascular disease
3. Having surgery other than oncological surgery
4. having coagulation disorder
5. being illiterate
6. having visual and auditory problems
7. Inability to cooperate with cognitive function test
8. having an emergency surgery
9. Those who are not able to read and sign the consent form
10. Patients deemed unsuitable by the researcher
11. Patients who do not want to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who will undergo major abdominoplasty, ASA II and ASA III, over the age of 18, under the age of 85 in the Ankara Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Cognitive functions | postoperative day 3
  Cognitive functions will be evaluated with Mini-mental test in each patient on postoperative day 3.

SECONDARY OUTCOMES:
postoperative pain scores | 24 hours postoperatively
  Postoperative pain scores will be recorded. The evaluation will be made with Visual Analogue Scale (VAS) score in the 1st, 2nd, 6th, 12th and 24th hours postoperatively.
  VAS score is determined via using a ruler, measuring the distance on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10.
Postoperative morphine consumption within 24 hours postoperatively | 24 hours postoperatively
  Total morphine consumption in 24 hours postoperatively will be recorded via Patient Controlled Analgesi (PCA) device.

CONTACTS AND LOCATIONS:
Overall Officials: Guldeniz Argun, 1, Study Chair — SBU Abdurrahman YAOTRH
Locations (1):
- SBU Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krenk L, Rasmussen LS, Kehlet H. New insights into the pathophysiology of postoperative cognitive dysfunction. Acta Anaesthesiol Scand. 2010 Sep;54(8):951-6. doi: 10.1111/j.1399-6576.2010.02268.x. Epub 2010 Jul 12. PMID 20626359
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Yirmiya R, Goshen I. Immune modulation of learning, memory, neural plasticity and neurogenesis. Brain Behav Immun. 2011 Feb;25(2):181-213. doi: 10.1016/j.bbi.2010.10.015. Epub 2010 Oct 21. PMID 20970492
- [Result] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Result] Statzer N, Cummings KC 3rd. Transversus Abdominis Plane Blocks. Adv Anesth. 2018 Dec;36(1):163-180. doi: 10.1016/j.aan.2018.07.007. Epub 2018 Sep 27. No abstract available. PMID 30414636
- [Result] Tulgar S, Ahiskalioglu A, Selvi O, Thomas DT, Ozer Z. Similarities between external oblique fascial plane block and blockage of thoracoabdominal nerves through perichondral approach (TAPA). J Clin Anesth. 2019 Nov;57:91-92. doi: 10.1016/j.jclinane.2019.03.027. Epub 2019 Mar 29. No abstract available. PMID 30933854
- [Result] Ohgoshi Y, Ando A, Kawamata N, Kubo EN. Continuous modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) for major abdominal surgery. J Clin Anesth. 2020 Mar;60:45-46. doi: 10.1016/j.jclinane.2019.08.031. Epub 2019 Aug 20. No abstract available. PMID 31442859